CLINICAL TRIAL: NCT01435369
Title: Phase II Study to Evaluate the Safety, Tolerability and Efficacy of CT-011 Administered Intravenously to Patients With Metastatic Melanoma
Brief Title: Safety, Tolerability and Efficacy Study of the Monoclonal Antibody, CT-011, in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-2011-01; 2011-004501-24 (EudraCT Number)
Record Dates: First submitted 2011-09-08; First posted 2011-09-16 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Melanoma; Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — pidilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT-011 at dose level 1 (1.5 mg/kg). (Active Comparator)
  Interventions: Drug: CT-011
- CT-011 at dose level 2 (6 mg/kg). (Active Comparator)
  Interventions: Drug: CT-011

INTERVENTIONS:
Drug: CT-011 — The monoclonal antibody, CT-011 is administered intravenously at 2 dosage levels, 1.5mg/kg and 6.0 mg/kg to patients with metastatic melanoma. The study drug will be given every other week for a total of up to 27 study drug infusions for about 12 months.

SUMMARY:
The purpose of this research study is to see if the study drug, CT-011, is safe to give and if it helps people with melanoma that has spread to other areas of their body. CT-011 is a monoclonal antibody. Monoclonal antibodies are a type of drug that is typically given by infusion into a vein (intravenously). Monoclonal antibodies are antibodies made in a lab instead of by the immune system which then recruit the immune system to help fight cancer cells.

All final eligible subjects will receive an intravenous infusion of CT-011. This study will test two dose levels of the study drug:

Group 1: Patients in this group will be given the study drug at dose level 1 (1.5 mg/kg).

Group 2: Patients in this group will be given the study drug at dose level 2 (6.0 mg/kg).

Each group will be given the study drug through an IV (a needle put into a vein in the arm) on day 1. After day 1, the study drug will be given every other week. Patients may be given a total of up to 27 study drug infusions for about 12 months while they are in the study. Approximately 100 patients will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a histologically or cytologically documented diagnosis of metastatic melanoma.
2. Participants age is 18 years or older.
3. Stage IV disease that is clearly progressive since last therapy
4. ECOG performance status of 0 or 1.

Exclusion Criteria:

1. Patients with uveal melanoma.
2. Active autoimmune disease, symptoms or conditions except for vitiligo, type I diabetes, treated thyroiditis, asymptomatic laboratory evidence of autoimmune disease (eg: + ANA, +RF, antithyroglobulin antibodies) or mild arthritis requiring no therapy or manageable with NSAIDs.
3. Prior use of anti PD-1, anti PD-L1 or PD-L2 therapy.
4. More than 3 prior lines of treatment for metastatic melanoma including approved and investigational treatments.
5. Women of child bearing potential who are pregnant

Note: This is only a partial list of eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The objective response rate (ORR) by Immune Related Response Criteria (irRC) in patients with metastatic melanoma treated with CT-011 | Approximately 28 months

SECONDARY OUTCOMES:
Safety of CT-011 | Approximately 28 months
  Safety will be assessed for incidence of Adverse Events
Progression Free Survival by Immune Related Response Criteria | Approximately 28 months
Overall Survival | Approximately 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Atkins, M.D., Principal Investigator — Beth Israel Deaconess Cancer Center
Locations (18):
- United States (16):
  - Yale University School of Medicine, Section of Med Onc., New Haven, Connecticut
  - Moffitt Cancer Center Cutaneous Oncology Department, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Mass General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ruttenberg Cancer Clinic - The Mount Sinai Hospital, New York, New York
  - Providence Cancer Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Univesity Medical Center, Dallas, Texas
  - University of Virginia Health System / Human Immune Therapy Center, Charlottesville, Virginia
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Chaim Sheba Medical Center, Tel Litwinsky